CLINICAL TRIAL: NCT05906030
Title: Diaphragm Dysfunction and Respiratory Complications in the Perioperative Setting- Can Diaphragm Ultrasound Aid Prediction?
Brief Title: Diaphragm Dysfunction and Ultrasound Perioperatively
Acronym: DiaphPeriop
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jessica Kåhlin, Medical Doctor, PhD, Karolinska University Hospital
Other Study IDs: K2023-3473
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Insufficiency; Pneumonia; Desaturation of Blood; Tachypnea; Atelectasis, Postoperative
Keywords: Diaphragm dysfunction; Postoperative complication; Respiratory complication; Pneumonia; Respiratory insufficiency
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia; Tachypnea; Pulmonary Atelectasis; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Diaphragm ultrasound — Diaphragm ultrasound will be used pre- and postoperatively. Diaphragm dysfunction will be diagnosed using the measurements diaphragm thickening fraction, diaphragm excursion and diaphragm density.

SUMMARY:
This study aims at determining whether diaphragm ultrasound examining diaphragm thickening fraction, excursion and density before and after surgery can predict respiratory complications in the postoperative period.

Patients scheduled for major elective abdominal, pelvic or vascular surgery will be included in the study and diaphragm ultrasound is performed before surgery and after surgery in the postoperative ward. Physiological parameters, laboratory parameters, data on surgery and anesthesia and comorbidities will be registered. Complications such as pneumonia, desaturation, need for intubation and other respiratory events up to 30 days will be registered and later correlated with the diaphragm measurements.

DETAILED DESCRIPTION:
Background

A considerable part of the population undergo surgery every year and in Sweden around 600,000 surgeries are registered yearly. Occurring complications after surgery include wound infections, urinary tract infections, venous thromboembolism and pneumonia. Postoperative pneumonia is the third most common complication and increases morbidity and mortality substantially(1). Furthermore, it prolongs hospital length of stay (LOS), increases medical costs and hospital readmissions. The incidence of postoperative pneumonia is dependent on non-modifiable factors such as type of surgery, age, sex and preoperative functional status but also on modifiable factors like smoking and adherence to preventive bundles(2). However, pneumonia preventive bundles are more studied and used in the ICU than in the perioperative setting. The current burden of postoperative pneumonia in Sweden is presently unknown. Furthermore, few prognostic examinations and preventive measures are used in the perioperative setting. It is well known that diaphragm dysfunction affects patients after major abdominal surgery and that it affects outcome postoperatively(3, 4). The mechanism behind the diaphragm dysfunction is unclear but animal studies indicate that postoperative inflammation may weaken the diaphragm only hours after exposure(5). Postoperative respiratory complications are partly due to a deteriorated diaphragm function and cause increased morbidity and mortality(6). In cardiac and upper abdominal surgery patients, ultrasound measurements of diaphragm excursion and thickening proved useful in ruling out diaphragm dysfunction(7, 8).

Diaphragm dysfunction can be diagnosed using ultrasound measuring diaphragm excursion, diaphragm thickness, thickening or diaphragm density. The examinations have high intra- and inter-observer reliability, are non-invasive and non-ionizing imaging techniques. This is in sharp contrast to twitch magnetic phrenic nerve stimulation, the golden standard technique for measuring diaphragm function, being reliable but invasive(9). Electric impedance tomography (EIT) is a non-invasive radiation-free imaging technique that provides real-time images and data of regional lung ventilation and lung volumes (10) and the correlation to diaphragm dysfunction and the later development of atelectases as assessed with ultrasound of the diaphragm is not clear. Furthermore, parameters on lung volumes retrieve with spirometry also lack a clear relationship with diaphragm ultrasound parameters and later respiratory complications.

Diaphragm ultrasound has previously been used to identify severe dysfunction. However, to identify early signs of dysfunction could render important actions perioperatively to avoid progression and continuation of early diaphragm dysfunction and hence an increased risk of complications.

Gap of knowledge Can diaphragm ultrasound in the peroperative setting predict respiratory complication after dismissal from postoperative ward? And can diaphragm dysfunction as defined with ultrasound be correlated to changes in lung volumes and lung function as demonstrated with EIT and spirometry?

Hypothesis We hypothesize that diaphragm ultrasound parameters indicating diaphragm dysfunction can predict respiratory complications in the perioperative setting.

Aims Overall aim To perform a comprehensive mapping of respiratory complications in the perioperative setting and to determine whether diaphragm dysfunction determined with diaphragm ultrasound can aid in predicting respiratory complications after major surgery.

Specific aims

1. To determine whether attenuated diaphragm function measured with diaphragm ultrasound before and after major elective abdominal, pelvic or vascular surgery can predict respiratory complications at 30 days.
2. To determine whether attenuated diaphragm function measured with diaphragm ultrasound before and after major acute abdominal, pelvic or vascular surgery can predict respiratory complications at 30 days.

Primary endpoint Pneumonia in the first postoperative week in relation to reduced diaphragm function.

Secondary endpoints Desaturation <90% in the postoperative ward or in the ward, takypnea >30 breaths/minute in the postoperative ward or in the ward, PaO2<9 in the postoperative ward, PaCO2>7 in the postoperative ward, need for intubation, need for non-invasive ventilation (NIV).

Design of study Prospective non-randomized observational study

Inclusion criteria

1. Adult, ≥18 years old
2. Planned for elective (study 1) or acute (study 2) abdominal, vascular or pelvic surgery at Karolinska University Hospital, Solna during the study period

Exclusion criteria

1. Chronic lung disease
2. Patients incapable of giving consent
3. Pregnancy

Methods

Patients 18 years and older undergoing open abdominal, pelvic or vascular surgery at the Karolinska University Hospital will be examined with diaphragm ultrasound measuring diaphragm excursion, thickness and density before surgery and before discharge from the postoperative ward. Respiratory complications up to 30 days after surgery will be recorded from the patients´ charts and correlated with the ultrasound parameters.

1. In a first study elective abdominal, pelvic or vascular surgery patients will be examined with diaphragm ultrasound preoperatively and (2-3 times) at the postoperative unit. The patients will be observed at the ward with regards to pulseoximetry, need for oxygen, vital parameters etc. These parameters will be correlated with registered respiratory complications at 30 days.
2. In a second study, acute abdominal, pelvic or vascular surgery patients will be examined with diaphragm ultrasound, preoperatively (on the operating table before anesthesia) and (2-3 times) at the postoperative unit and subsequently observed at the ward with regards to pulseoximetry, need for oxygen, vital parameters etc. Retrieved parameters will be correlated with registered respiratory complications at 30 days.

Prior to these studies the method will be validated according to standards.

The examination of the diaphragm will be performed with the ultrasound machines normally used at the units. A curved transducer with the frequency 2,5-3,5 MHz or a linear transducer with the frequency 7,5-10 MHz is placed in the supine position at the right and left costal arch measuring the movement of the diaphragm at inspiration, the thickening of the diaphragm at inspiration and the diaphragm density. The examination is pain-free, non-invasive, non-radiating and takes about 15 minutes.

1. Diaphragm excursion:

   The movement of the diaphragm at inspiration is measured with a convex/curved transducer. On the right side, the probe is placed between the mid-clavicular line and the anterior axillary line under the costal arch. The probe is angled medially, cranially and dorsally to hit the diaphragm cupola in a perpendicular manner. The displacement of the diaphragm with inspiration is measured and registered in M-mode.
2. To measure diaphragm thickening the probe is placed between the 8:th and 9:th rib between the antero- and midaxillary line. The right diaphragm curvature is found 0,5-2 cm beneath the phrenicocostal sinus. M-mode is used to measure the thickness from the pleural line to the peritoneal line at forced residual capacity (FRC) and total lung capacity (TLC), I e at maximal inspiration. Normal thickening is 2,7mm +-0.5 mm and values under 2mm (<20%) are considered pathological.
3. Diaphragm density is measured in B-mode whereby a grayscale histogram is created with a special software (Image J or similar). The density is measured in percent of a grayscale where a value >65% (based on grayscale histograms on healthy controls) is defined as pathological.

The examination of the diaphragm will be performed pre-operatively on the operating ward. Postoperatively, the patient is examined on the operating table if possible and at two more occasions on the postoperative ward.

On the postoperative ward, the patient's vital functions are monitored and this data will be registered in the CRF (saturation, pulse, blood pressure, breathing frequency, pain estimation). Data on medications, anesthetics, surgery time, anesthesia time, perioperative bleeding, fluid balance, When the patient is transferred to the ward, a member of the research group will perform a follow-up ultrasound 24-72h after the first ultrasound. At this timepoint, vital parameters, data on medications, fluid balance and complications will be registered.

The patient will thereafter be followed up in Take Care (and Clinisoft if admitted to the ICU) with regards to respiratory complications up to 30 days after the initial surgery.

Data from the diaphragm ultrasounds will be saved in the ultrasound machine and exported as both pictures and numerical files to pass word-protected hard disks.

Statistics Comparison of the primary outcome will be analysed with the Pearson chi-square test or two-tailed Fisher exact test for each diaphragm parameter. Baseline patient characteristic data will be described, and secondary outcomes, as described above, will be analysed as appropriate, depending on categorical or continuous parameters and normal or non-normal distribution. Data will be presented as mean ± SD or 95% CI, as median and range or numbers (%) dependent on the above.

Clinical relevance

This project will perform a unique mapping of the magnitude of postoperative complications after major surgery in Sweden. Several studies demonstrate diaphragm weakness after major surgery which predisposes the patient to respiratory complications postoperatively. Early detection of diaphragm weakness in the perioperative setting would give an opportunity to prevent respiratory complications by introducing pneumonia bundles, physiotherapy and increase awareness of symptoms of complications. Postoperative respiratory complications impose great challenges on the individual´s recovery as well as on health care costs. To introduce a non-invasive, reliable, cheap and painless diagnostic tool that could aid in the prevention of such complications would reduce both burden of illness and costs related to surgery.

References

1. Kazaure HS, Martin M, Yoon JK, Wren SM. Long-term results of a postoperative pneumonia prevention program for the inpatient surgical ward. JAMA Surg. 2014;149(9):914-8.
2. Chughtai M, Gwam CU, Mohamed N, Khlopas A, Newman JM, Khan R, et al. The Epidemiology and Risk Factors for Postoperative Pneumonia. J Clin Med Res. 2017;9(6):466-75.
3. Ford GT, Whitelaw WA, Rosenal TW, Cruse PJ, Guenter CA. Diaphragm function after upper abdominal surgery in humans. The American review of respiratory disease. 1983;127(4):431-6.
4. Berdah SV, Picaud R, Jammes Y. Surface diaphragmatic electromyogram changes after laparotomy. Clin Physiol Funct Imaging. 2002;22(2):157-60.
5. Krause KM, Moody MR, Andrade FH, Taylor AA, Miller CC, 3rd, Kobzik L, et al. Peritonitis causes diaphragm weakness in rats. Am J Respir Crit Care Med. 1998;157(4 Pt 1):1277-82.
6. Sasaki N, Meyer MJ, Eikermann M. Postoperative respiratory muscle dysfunction: pathophysiology and preventive strategies. Anesthesiology. 2013;118(4):961-78.
7. Lerolle N, Guérot E, Dimassi S, Zegdi R, Faisy C, Fagon JY, et al. Ultrasonographic diagnostic criterion for severe diaphragmatic dysfunction after cardiac surgery. Chest. 2009;135(2):401-7.
8. Kim SH, Na S, Choi JS, Na SH, Shin S, Koh SO. An evaluation of diaphragmatic movement by M-mode sonography as a predictor of pulmonary dysfunction after upper abdominal surgery. Anesth Analg. 2010;110(5):1349-54.
9. Doorduin J, van Hees HW, van der Hoeven JG, Heunks LM. Monitoring of the respiratory muscles in the critically ill. Am J Respir Crit Care Med. 2013;187(1):20-7.
10. Lobo B, Hermosa C, Abella A, Gordo F. Electrical impedance tomography. Ann Transl Med. 2018;6(2):26.

ELIGIBILITY:
Inclusion Criteria:

Adults undergoing elective (study 1) or acute (study 2) abdominal, pelvic or vascular surgery

Exclusion Criteria:

* <18 years
* Underlying chronic respiratory disease
* Patients not able to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing elective (study 1) or acute (study 2) abdominal, pelvic or vascular surgery
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Pneumonia | 30 days
Respiratory insufficiency | 30 days
  Need for non-invasive or invasive ventilation
Desaturation | 30 days
  Need for supplemental oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kåhlin, Principal Investigator — Karolinska Universitetssjukhuset Solna
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Perioperative Medicine and Intensive Care, Stockholm, Stockholm County
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No
IPD may be shared upon request